CLINICAL TRIAL: NCT06321848
Title: The Predictive Value Of Heart, Lung And Diaphragm Ultrasound For Ventilator Weaning Outcome Of Surgical Intensive Care Patients
Brief Title: Weaning Ventilator Using Heart, Lung And Diaphragm Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: DUCGM2426
Record Dates: First submitted 2024-02-27; First posted 2024-03-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Ventilator Weaning; Ultrasound
Keywords: echocardiography; lung ultrasound; diaphragm ultrasound; ventilator weaning

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The ventilator weaning patients: Patients who have been on mechanical breathing for longer than 48 hours using an endotracheal tube and who fit the requirements to be weaned off of it

SUMMARY:
Postextubation distress is detrimental to the prognosis of critically ill patients with successful spontaneous breathing trial. Failure to wean is known to be connected with heart, lung, and diaphragm problems. The aim of this study was to investigate how a composite model comprising diaphragm, lung, and heart ultrasonography indications could predict the weaning outcome.

Methods: Ultrasonic features of the diaphragm, heart, and lungs are going to be collected along with clinical data about the patients. Either the successful weaning group or the failed weaning group is going to comprised the patients. Multivariate logistic regression analysis is going to be used to identify the variables that may be associated with the likelihood of weaning failure. A multiindicator combination model is going to be developed to increase the predictive accuracy after the possible indicators' accuracy in foretelling the weaning outcome was assessed.

DETAILED DESCRIPTION:
- Research participants: From March 2024 to March 2026 in the Department of Anesthesia, critical care and pain medicine, Hanoi Medical University Hospital, patients ages over 18 years who will have mechanically ventilated for over 48 h will be recruited. Patients will be excluded if they had a diagnosis of progressive neuromuscular diseases, a history of cardiovascular or respiratory disease who depend on a ventilator at home (COPD, severe bronchial asthma), patients with thoracic surgery and mitral valve surgery. All patients and their families signed informed consents.

- Clinical data collection: Clinical data including gender, age, body mass index, primary disease, length of stay in ICU, duration of mechanical ventilation, acute physiology and chronic health evaluation II, Charlson Comorbidity Index, history of surgery/internal diseases will be collected.

- Spontaneous breathing trial (SBT): Patients will be undergone a 60-min SBT when they meet all the readiness weaning criteria with PS 7cmH2O, PEEP 5cmH2O, FiO2 40%. The vital signs, rapid shallow breathing index (RSBI), NIF, P0.1, tidal volume, respiratory rate, arterial blood gases will be recorded at the beginning and at the end of SBT.

GE Logiq P7 (GE Healthcare, USA) and Philips Affiniti 70G (Philips Ultrasound, USA) ultrasound diagnostic instruments will be used in this study. The heart, lung and diagphragm ultrasonic findings will be recorded by the sonographer well trained in point-of-care ultrasound at the begining and at the end of the SBT.

Tracheal extubation is carried out if the patient does not exhibit symptoms of intolerance, indicating that the SBT treatment was successful. In case intolerance symptoms manifest, return to the initially chosen breathing mode (SIMV, A/C) and record the SBT failure.

- Extubation: After successful SBT: proceed with extubation. The patient is given an oxygen mask at 5L/minute. If the patient does not show intolerance symptoms within 48 hours, the extubation is considered successful. If the patient develops one of the intolerance symptoms during this time period, the extubation failure will be recorded and the patients will be reintubated. Record the values of vital signs and arterial blood gas variables every 24, 48 hours after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* The duration of postoperative mechanical ventilation >= 48 hours

Exclusion Criteria:

* Patient had a diagnosis of progressive neuromuscular diseases
* Patient had a history of cardiovascular or respiratory disease who depend on a ventilator at home (COPD, severe bronchial asthma)
* Patients had thoracic surgery or mitral valve surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a duration of mechanical ventilation through an endotracheal tube of more than 48 hours and meeting the criteria of readiness to wean off mechanical ventilation will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The ventilator weaning outcome | after 48 hours of extubation
  The outcome of weaning ventilation process (successful or failure)

SECONDARY OUTCOMES:
The hospital length of stay | Approximately 5-15 days postextubation
  The time between hospital admission and discharge
The ICU length of stay | Approximately 2-15 days postextubation
  The time between ICU admission and discharge
The duration of mechanical ventilation | Daily assessment of requirement of mechanical ventilation from the time of intubation until the date of weaning mechanical ventilation, up to 12 months
  The time from the start of mechanical ventilation to extubation

CONTACTS AND LOCATIONS:
Overall Officials: Tu Nguyen, Professor, Study Director — Hanoi Medical University
Locations (1):
- Hanoi Medical University Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The investigators agree that all results and conclusion of this research will be used fully for other researchers
Supporting Information: Study Protocol, ICF, CSR
Time Frame: from March 2026 to the unidentified time
Access Criteria: anesthesiologists all over the world